CLINICAL TRIAL: NCT04037059
Title: Impact of Body Habitus (Arm Span and Abdominal Girth) on Activities of Daily Living (ADL) in Patients Undergoing Long Segment Deformity Surgery: A Prospective Study
Brief Title: Impact of Body Habitus (Arm Span and Abdominal Girth) on Activities of Daily Living (ADL)
Acronym: ADL
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00101177
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2021-10

CONDITIONS: Spinal Fusion; Activities of Daily Living Following Complex Spinal Fusions
Keywords: Activities of Daily Living (ADL); Complex Spinal Fusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal Deformity Patients: For patients with disabling spinal deformities, long segment fusions have been shown to improve the health related quality of life (HRQOL). A consequence of spine fusion however is elimination of range of motion especially in the lumbar spine. Even in patients who report overall improvement in pain related domains, difficulty with some ADL's in this patient group has been well documented in previous studies. Complaints such as inability to dress independently, bathing of lower halves of their body, driving a motor vehicle, getting in and out of a chair/bed and performing perineal hygiene care following toileting have been reported.

SUMMARY:
This study is being done to assess the impact of arm length and abdominal (belly) width on patient performance of daily self-care activities following multiple level spinal fusions. The study will also assess if the number of levels operated on in the spinal fusion procedure affects your ability to perform Activities of Daily Living (ADL) and how long after surgery do the difficulties/limitations persist.

DETAILED DESCRIPTION:
This is a prospective, single-center study of adult patients undergoing long segment spinal fusions to the pelvis (>5 levels).

Health Related Quality of Life Outcome (HRQOL) consisting of the Oswestry Disability Index (ODI), Visual Analog Scale, EQ-5D, Scoliosis Research Society-22 and 30 (SRS-22 and SRS-30) and the Lumbar Stiffness Disability Index (LSDI) will be collected preoperatively, 6 weeks, 3 months, 6 months, 12 and 24 months. All measures will be collected during clinic visits.

Primary and secondary objectives The primary objective is to determine the impact of body habitus on postoperative ADLs in patients undergoing long segment spinal fusions.

The secondary objective will be to determine if the number of levels of fusions impact the ability to perform ADLs and to study how long after surgery do the difficulties/limitations persist.

Study procedures Enrolled subjects meeting eligibility criteria and provide consent will be approached by the study coordinator and explained the purpose of the study, risks and benefits to participation, and queried about their interest in participation. Patients consenting to the study will have the following measurements performed by the clinician with an evaluation prior to surgery, during their 6 week, 3 month, 6 month, 12 and 24 month postoperative visits.

1. Waist circumference using a measuring tape will be obtained from midway between the last ribs and the iliac crest as suggested by the World Health Organization and the International Diabetes Federation.
2. The arm span (wingspan) or reach will be measured. To measure the arm span, the patient will be asked to stand against the wall with their arms extended sideways at a ninety-degree angle. Using a measuring tape, the distance from the tip of the middle finger of one hand to the tip of the middle finger in other arm will be measured and recorded.
3. The distance from the ground to the tip of middle finger will be measured while the patient is asked to touch their toes with knees fully extended.

As mentioned, all study patients will complete Health Related Quality of Life Outcome (HRQOL) consisting Oswestry Disability Index (ODI), Visual Analog Scale, EQ-5D, Scoliosis Research Society-22 (SRS-22) and the Lumbar Stiffness Disability Index (LSDI) at 6 weeks, 3 months, 6 month, 12 and 24 months.

Data will be collected in a password-protected file and will be stored in an electronically secure environment, as specified in the research data security plan (RDSP).

Follow-up by the research coordinator as part of this study will not necessarily preclude or replace any follow-up by the treating physician or nursing staff as part of the routine standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Adults18 to 80 years old
2. Spinal fusion surgery involving thoracolumbar spine > 5 levels
3. Ability to stand to obtain arm span, abdominal girth and ability to bend at the waist to obtain measurement

Exclusion Criteria:

1. Patients who are incarcerated, paraplegic or unable to return for follow-up visits
2. Patients with prior lumbar fusions at the indicated levels for surgery
3. Spinal fusion surgery involving thoracolumbar < 5 levels
4. Patients who already have lumbopelvic fixation with iliac screws

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are seeking evaluation and treatment at the Duke Spine Center and have been recommended to undergo spine surgery will be approached by the treating surgeon and/or the study coordinator about the study.
  The goal enrollment is 256 patients within 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life as measured by Oswestry Disability Index (ODI) | Baseline, 6 weeks, 3 months, 6 months, 12 and 24 months
  10 question survey that rates disability from low, moderate, to severe disability
Change in Quality of Life as measured by Visual Analog Scale (VAS) | Baseline, 6 weeks, 3 months, 6 months, 12 and 24 months
  4 question survey that rates pain
Change in Quality of Life as measured by EQ-5D | Baseline, 6 weeks, 3 months, 6 months, 12 and 24 months
  Survey that looks at 5 different components activities of daily living
Change in Quality of Life as measured by Scoliosis Research Society (SRS) Form | Baseline, 6 weeks, 3 months, 6 months, 12 and 24 months
  22 or 30 question survey that rates scoliosis
Change in Quality of Life as measured by Lumbar Stiffness Disability Index (LSDI) Form | Baseline, 6 weeks, 3 months, 6 months, 12 and 24 months
  Survey that rates lumbar stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Karikari, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No